CLINICAL TRIAL: NCT02103556
Title: Double-blind Randomized Trial on the Effect of Olive Oil and Flaxseed Oil on Constipation of Hemodialysis Patients
Brief Title: Edible Oils in the Treatment of Constipation of Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Lilian Cuppari, Affiliate Professor, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2012/06605-9
Record Dates: First submitted 2014-03-10; First posted 2014-04-04 (Estimated); Last update posted 2014-04-04 (Estimated); Status verified 2014-04

CONDITIONS: Chronic Kidney Disease
Keywords: Constipation; Rome III criteria; Hemodialysis
MeSH Terms: conditions — Renal Insufficiency, Chronic; Constipation | interventions — Mineral Oil; Olive Oil; Linseed Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Mineral oil (Active Comparator): 4ml daily (adjusted as needed), for 4 weeks
  Interventions: Other: Mineral oil
- Olive oil (Active Comparator): 4ml daily (adjusted as needed), for 4 weeks
  Interventions: Dietary Supplement: Olive oil
- Flaxseed oil (Active Comparator): 4 ml daily (adjusted as needed), for 4 weeks
  Interventions: Dietary Supplement: Flaxseed oil

INTERVENTIONS:
Other: Mineral oil — 4 ml daily (adjusted as needed), for 4 weeks
  Arms: Mineral oil
Dietary Supplement: Olive oil — 4 ml daily (adjusted as needed), for 4 weeks
  Arms: Olive oil
Dietary Supplement: Flaxseed oil — 4 ml daily (adjusted as needed), for 4 weeks
  Arms: Flaxseed oil

SUMMARY:
The purpose of this study was to evaluate the effect of olive oil and flaxseed oil in the treatment of constipation of patients undergoing hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

* Constipated patients by Rome III criteria
* Hemodialysis > 3 months

Exclusion Criteria:

* Diagnosis of gastrointestinal disease other than constipation
* Previous intolerance to the oils used in the study
* Cognitive limitations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-04; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Score of constipation symptoms | 1 month
  Constipation was diagnosed by the Rome III criterion. The diagnosis consists in the presence, for at least three months, of two or more of the following symptoms: "fewer than three evacuations per week", "straining on evacuation", "lumpy or hard stools", "incomplete evacuation", "anorectal obstruction" and use of "manual maneuvers" to facilitate evacuation. Each symptom is scored as: 0=never or rarely, 1=sometimes, 2=often, 3=most of the time and 4=always. In the present study, the frequency of the symptoms was considered as a continuous variable and, a final score ranging from 0 to 24 was calculated. Lowest scores were indicative of fewer symptoms of constipation.

CONTACTS AND LOCATIONS:
Overall Officials: Lilian Cuppari, PhD, Principal Investigator — Federal University of São Paulo; Christiane I Ramos, Principal Investigator — Federal University of São Paulo
Locations (1):
- Federal University of São Paulo, São Paulo, São Paulo, Brazil